CLINICAL TRIAL: NCT00158847
Title: Modification of Disease Outcome in COPD. Shortterm Versus Longterm Treatment With Inhaled Corticosteroids, Either or Not Combined With a Long-Acting Beta2-Agonist.
Brief Title: Modification Of Disease Outcome In COPD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Academisch Ziekenhuis Groningen (Other); The Netherlands Asthma Foundation (Other); Netherlands Organisation for Scientific Research (Other Government); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO30001; SER9804 / Glucold
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-01-20 (Estimated); Status verified 2005-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD inflammation sputum lung function biopsy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate

INTERVENTIONS:
Drug: fluticasone 500 mcg
Drug: fluticasone 500 mcg + salmeterol 50 mcg

SUMMARY:
The hypothesis to be tested of this study is that treatment with fluticasone propionate leads to an initial improvement in symptoms, quality of life and lungfunction and a reduction in airways hyperresponsiveness. The continued decline of lungfunction in COPD may not be influenced by longer lasting treatment. Addition of salmeterol will augment the initial benefits of fluticasone without changing the longterm decline in lungfunction.

DETAILED DESCRIPTION:
Aim The primary aim of this study was to investigate whether short-term treatment with inhaled corticosteroids in COPD results in greater improvements in airway pathology, thereby leading to larger clinical benefits, than continuous long-term treatment. To that end, the outcome variables included features of airways inflammation and remodelling as well as clinical symptoms, exacerbations, quality of life, decline in FEV1, bronchial responsiveness, and pharmaco-economics. The secondary aim of the study was to examine the histopathological and clinical benefits of the combined treatment with an inhaled steroid and a long-acting ß2-agonist in COPD.

Methods Patients. Patients with COPD (45-75 yr, >10 pckyr) not using inhaled steroids for the past 3 months were recruited.

Design. In a prospective, longitudinal, double blind, 4-arm study, the patients were followed during 2.5 years (Figure 1). They were treated with high dose inhaled corticosteroids (500 g fluticasone bid), combined inhaled steroids+long-acting ß2-agonist (500 µg fluticasone+50 µg salmeterol) or placebo for 6 months. Half of the patients in the steroid group continued their treatment with steroids for another 2 years, whereas the other half received placebo. The combination therapy and placebo groups remained unaltered treatment up to 2.5 years.

Measurements. Symptoms, exacerbations, QOL questionnaires and spirometry were monitored every 3 months. Peripheral blood eosinophils, IgE, exhaled NO, bodyplethysmography, CO-diffusion capacity, PC20 methacholine, sputum induction and bronchoscopy were performed at 0, 6, and 30 months. In BAL and induced sputum we are measuring cell differentials and their state of activation. Immunohistochemistry is being performed in bronchial biopsy specimens, staining for markers on infiltrative and resident cells, and morphometric analysis will allow airway remodelling to be quantified, by using a computerized image analysis system. The effects of treatment will be analyzed by relating the observed changes in clinical and pathophysiological outcome, to those in cellular and histological outcome by using linear mixed statistical models.

ELIGIBILITY:
Inclusion criteria:

* COPD patients with > 10 pack years.
* Written informed consent.
* Able to complete a diary card.
* At least one of the following symptoms: chronic cough, chronic sputum production, frequent exacerbations, or dyspnoea at exertion.
* Postbronchodilator FEV1 below 90% confidence interval of predicted and postbronchodilator FEV1/FVC below 90% confidence interval of predicted.

Exclusion criteria:

* No oral corticosteroids 3 months prior to the study or maintenance treatment with corticostroids 6 months prior to the study.
* No history of asthma, lung diseases other than COPD, other diseases likely to interfere with the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2000-04; Study Completion 2005-05

PRIMARY OUTCOMES:
Inflammation: localisation, numbers and profile of neutrophils, eosinophils, macrophages, and CD8+T cells in bronchial biopsy specimens after 6 months and 2.5 years treatment.

SECONDARY OUTCOMES:
Clinical: symptoms, exacerbations, quality of life, lung function, 6 min walking test. Inflammation: markers in sputum and BAL, profile of epithelial cells, remodeling.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Sterk, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden

REFERENCES:
- [Background] Lapperre TS, Snoeck-Stroband JB, Gosman MM, Stolk J, Sont JK, Jansen DF, Kerstjens HA, Postma DS, Sterk PJ; Groningen and Leiden Universities Corticosteroids in Obstructive Lung Disease Study Group. Dissociation of lung function and airway inflammation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Sep 1;170(5):499-504. doi: 10.1164/rccm.200401-112OC. Epub 2004 Jun 1. PMID 15172889
- [Derived] Fang J, Wolters JC, Rafie K, Wang C, Bartel S, van den Berge M, Hylkema MN. Extracellular vesicles from bronchoalveolar lavage fluid provide insights into the inhaled corticosteroids treatment response in COPD. Respir Res. 2025 Jul 30;26(1):254. doi: 10.1186/s12931-025-03330-6. PMID 40739568
- [Derived] Ditz B, Boekhoudt J, Couto N, Brandsma CA, Hiemstra PS, Tew GW, Neighbors M, Grimbaldeston MA, Timens W, Kerstjens HAM, Rossen JWA, Guryev V, van den Berge M, Faiz A. The Microbiome in Bronchial Biopsies from Smokers and Ex-Smokers with Stable COPD - A Metatranscriptomic Approach. COPD. 2022;19(1):81-87. doi: 10.1080/15412555.2022.2033193. Epub 2022 Feb 4. PMID 35118915
- [Derived] Faiz A, Imkamp K, van der Wiel E, Boudewijn IM, Koppelman GH, Brandsma CA, Kerstjens HAM, Timens W, Vroegop S, Pasma HR, Boersma WG, Wielders P, van den Elshout F, Mansour K, Steiling K, Spira A, Lenburg ME, Heijink IH, Postma DS, van den Berge M. Identifying a nasal gene expression signature associated with hyperinflation and treatment response in severe COPD. Sci Rep. 2020 Oct 15;10(1):17415. doi: 10.1038/s41598-020-72551-0. PMID 33060632
- [Derived] Kunz LI, van't Wout EF, van Schadewijk A, Postma DS, Kerstjens HA, Sterk PJ, Hiemstra PS. Regulation of YKL-40 expression by corticosteroids: effect on pro-inflammatory macrophages in vitro and its modulation in COPD in vivo. Respir Res. 2015 Dec 22;16:154. doi: 10.1186/s12931-015-0314-3. PMID 26696093
- [Derived] Snoeck-Stroband JB, Lapperre TS, Sterk PJ, Hiemstra PS, Thiadens HA, Boezen HM, Ten Hacken NH, Kerstjens HA, Postma DS, Timens W, Sont JK; GLUCOLD Study Group. Prediction of Long-Term Benefits of Inhaled Steroids by Phenotypic Markers in Moderate-to-Severe COPD: A Randomized Controlled Trial. PLoS One. 2015 Dec 10;10(12):e0143793. doi: 10.1371/journal.pone.0143793. eCollection 2015. PMID 26659582
- [Derived] Kunz LIZ, Postma DS, Klooster K, Lapperre TS, Vonk JM, Sont JK, Kerstjens HAM, Snoeck-Stroband JB, Hiemstra PS, Sterk PJ; GLUCOLD Study Group. Relapse in FEV1 Decline After Steroid Withdrawal in COPD. Chest. 2015 Aug;148(2):389-396. doi: 10.1378/chest.14-3091. PMID 25836351
- [Derived] Kunz LI, Strebus J, Budulac SE, Lapperre TS, Sterk PJ, Postma DS, Mauad T, Timens W, Hiemstra PS; GLUCOLD (Groningen Leiden Universities Corticosteroids in Obstructive Lung Disease) Study Group. Inhaled steroids modulate extracellular matrix composition in bronchial biopsies of COPD patients: a randomized, controlled trial. PLoS One. 2013 May 7;8(5):e63430. doi: 10.1371/journal.pone.0063430. Print 2013. PMID 23667615
- [Derived] Lapperre TS, Snoeck-Stroband JB, Gosman MM, Jansen DF, van Schadewijk A, Thiadens HA, Vonk JM, Boezen HM, Ten Hacken NH, Sont JK, Rabe KF, Kerstjens HA, Hiemstra PS, Timens W, Postma DS, Sterk PJ; Groningen Leiden Universities Corticosteroids in Obstructive Lung Disease Study Group. Effect of fluticasone with and without salmeterol on pulmonary outcomes in chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2009 Oct 20;151(8):517-27. doi: 10.7326/0003-4819-151-8-200910200-00004. PMID 19841453
- [Derived] Lapperre TS, Sont JK, van Schadewijk A, Gosman MM, Postma DS, Bajema IM, Timens W, Mauad T, Hiemstra PS; GLUCOLD Study Group. Smoking cessation and bronchial epithelial remodelling in COPD: a cross-sectional study. Respir Res. 2007 Nov 26;8(1):85. doi: 10.1186/1465-9921-8-85. PMID 18039368